CLINICAL TRIAL: NCT05453994
Title: Efficacy of Bismuth Added to Potassium-competitive Acid Blocker-based Triple Regimen for First-line Helicobacter Pylori Eradication
Brief Title: Bismuth for PCAB-based H. Pylori Eradication
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-HP-2022
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: H. Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-bismuth group: Tegoprazan 50 mg bid, amoxicillin 1000 mg bid, clarithromycin 500 mg bid for 14 days
  Interventions: Drug: H. pylori eradication
- Bismuth group: Tegoprazan 50 mg bid, amoxicillin 1000 mg bid, clarithromycin 500 mg bid, tripotassium dicitrate bismuthate (DENOL) 300 mg bid for 14 days
  Interventions: Drug: H. pylori eradication

INTERVENTIONS:
Drug: H. pylori eradication — PPIs-based Antimicrobial agents for H. pylori eradication

SUMMARY:
Tegoprazan is a new potassium-competitive acid blocker (PCAB) that has been clinically available since 2018 in South Korea. P-CAB is highly active drugs targeting H+, K+ -ATPase in the gastric acid secretion of parietal cells. The mechanism of action is different from that of PPIs. Conventional PPIs require 3-5 days to achieve maximal and steady-state gastric acid inhibition, whereas P-CAB increases the intragastric pH to nearly 7 within four hours. In Japan, H. pylori eradication success rates has increased by therapies using P-CAB than those using proton pump inhibitors, owing to the stronger acid suppression capability of P-CAB.

Bismuth has long been used to treat peptic ulcer disease, dyspepsia, parasite infections, and infectious diarrhea. The antibacterial effects of bismuth include inhibition of protein and cell wall synthesis in H. pylori. The main role of bismuth is to increase the eradication rate by 30%-40% in resistant H. pylori strains.

DETAILED DESCRIPTION:
The investigators aim to evaluate the success rate and adverse drug events of bismuth added to PCAB-based triple therapy as a first-line regimen for H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 80 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* Drug allergy to antibiotics
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: H. pylori-infected patients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
H. pylori infection status | 6 weeks
  Rate of successful H. pylori eradication

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Digestive Disease Center, Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JH. Bismuth add-on improves the efficacy of 2-week tegoprazan-based triple therapy for first-line Helicobacter pylori eradication: a real-world evidence study. Expert Rev Anti Infect Ther. 2024 Sep;22(9):793-799. doi: 10.1080/14787210.2024.2329251. Epub 2024 Mar 13. PMID 38459869